CLINICAL TRIAL: NCT03168438
Title: Open-Label Pilot Study to Assess the Safety, Tolerability and Antitumor Activity of Genetically Engineered NY-ESO-1 Specific (c259) T Cells Alone or in Combination With Pembrolizumab in HLA-A2+ Subjects With NY-ESO-1 and/or LAGE-1a Positive Relapsed and Refractory Multiple Myeloma
Brief Title: Letetresgene Autoleucel Engineered T Cells Alone and in Combination With Pembrolizumab in NY-ESO-1 Positive Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated following an internal review of the company's research and development portfolio
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 208470; ADP-0011-008 (Other: Adaptimmune Therapeutics); KEYNOTE-487 (Other: Merck Sharp and Dohme Corp.)
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-10

CONDITIONS: Neoplasms
Keywords: Relapsed and Refractory Multiple Myeloma; T Cell Receptor; Immuno-oncology; NY-ESO-1; Leukapheresis; Adoptive TCR T-cell therapy; Letetresgene autoleucel
MeSH Terms: conditions — Neoplasms; Recurrence; Multiple Myeloma | interventions — pembrolizumab; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Letetresgene autoleucel (GSK3377794) (Experimental): Eligible participants will be leukapheresed to manufacture engineered T-cells. Participants will then receive letetresgene autoleucel (GSK3377794), as a single intravenous (IV) infusion after completing lymphodepleting chemotherapy.
  Interventions: Drug: Letetresgene autoleucel; Drug: Fludarabine; Drug: Cyclophosphamide
- Arm 2: Letetresgene autoleucel (GSK3377794) with pembrolizumab (Experimental): Eligible participants will be leukapheresed to manufacture engineered T-cells. Participants will then receive letetresgene autoleucel (GSK3377794), as a single intravenous (IV) infusion after completing lymphodepleting chemotherapy, followed by pembrolizumab 200 mg every 3 weeks.
  Interventions: Drug: Letetresgene autoleucel with pembrolizumab; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Letetresgene autoleucel — Letetresgene autoleucel (GSK3377794) as an IV infusion
  Arms: Arm 1: Letetresgene autoleucel (GSK3377794)
Drug: Letetresgene autoleucel with pembrolizumab — Letetresgene autoleucel (GSK3377794) as an IV infusion, followed by pembrolizumab every 3 weeks
  Arms: Arm 2: Letetresgene autoleucel (GSK3377794) with pembrolizumab
Drug: Fludarabine — Fludarabine will be used as lymphodepleting chemotherapy and will be administered via IV route.
Drug: Cyclophosphamide — Cyclophosphamide will be used as lymphodepleting chemotherapy and will be administered via IV route.
Drug: Pembrolizumab — Pembrolizumab is available as an IV infusion
  Arms: Arm 2: Letetresgene autoleucel (GSK3377794) with pembrolizumab

SUMMARY:
This trial will evaluate safety, tolerability, and efficacy of letetresgene autoleucel (GSK3377794) with or without pembrolizumab in participants with relapsed and refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years of age or older on the date of signing informed consent.
* Histologically confirmed diagnosis of secretory multiple myeloma with myeloma markers at levels defined in the protocol.
* Documented diagnosis of relapsed and refractory multiple myeloma (RRMM) (at least 3 prior regimens and responsive to at least 1, and refractory to most recent prior therapies, which must have included one or more than one drug from each of the following drug classes: an immunomodulatory imide drug (IMiD), proteasome inhibitor, alkylator (unless the participant is ineligible or contraindicated to receive an alkylator), CD 38 monoclonal antibody, and glucocorticoid as separate lines or a combined line of therapy.- Left ventricular ejection fraction (LVEF) >= 50%. Lower LVEF (>= 40%) permissible if formal cardiologic evaluation reveals no evidence for clinically significant functional impairment.
* Meets protocol criteria for patients who have previously received checkpoint inhibitors or other immuno-oncology agents.
* ECOG Performance Status 0 or 1.
* Participant is HLA-A*02:01, HLA-A*02:05, and/or HLA-A*02:06 positive as determined by a designated central laboratory.
* Participant has confirmed sufficient expression of NY-ESO-1 and/or LAGE-1a as determined by a designated central laboratory.
* In the Investigator's opinion, the participant is fit for cell collection.
* Participant has adequate organ function and cell counts as described in the protocol.
* Participants previously treated with BCMA therapy (BCMA chimeric antigen receptor (CAR)-T, antibody-drug conjugate (ADC), or other type of BCMA-targeted therapy) must have progressed from this therapy prior to attending the Baseline visit prior to beginning lymphodepletion.
* Contraception use by male and female participant meets protocol requirements.

Exclusion Criteria:

* Has only plasmacytomas, plasma cell leukemia, monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), non-secretory myeloma or primarily amyloidosis.
* Previously received anti- programmed death (PD)-1, anti-PD-ligand (L)1, or anti-PD-L2 inhibitor.
* Previously participated in Merck pivotal trial NCT02576977: Study of Pomalidomide and Low Dose Dexamethasone With or Without Pembrolizumab in Refractory or RRMM.
* Had a prior allogeneic stem cell transplant.
* Has ongoing toxicity from previous anticancer therapy.
* Had a major surgery within 4 weeks prior to enrollment.
* Has history of allergic reactions to fludarabine, cyclophosphamide or agents similar to fludarabine, cyclophosphamide or other agents used in the study.
* Known history of myelodysplasia.
* Current active liver or biliary disease.
* Known history of chronic active hepatitis or liver cirrhosis.
* Participant has an active viral infection.
* History of severe immune disease, including non-infectious pneumonitis, requiring steroids or other immunosuppressive treatments.
* Active immune-mediated diseases.
* Prior or active demyelinating disease.
* Evidence or history of significant cardiac disease.
* Evidence or history of other significant, hepatic, renal, ophthalmologic, psychiatric, or gastrointestinal disease.
* Participants with concomitant second malignancies (except adequately treated non-melanomatous skin cancers, carcinoma in situ of the breast, treated superficial bladder cancer or prostate cancer, or in situ cervical cancers ) not in complete remission.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may be eligible.
* Active bacterial or systemic viral or fungal infections.
* Pregnant or breastfeeding.
* Cannot meet washout periods for prior radiotherapy, chemotherapy or other protocol-specified therapies.
* More than 2 years have passed since the participant's last leukapheresis collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (5):
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Nishihori T, Hoffman JE, Huff A, Kapoor GS, Eleftheriadou I, Zajic S, Urbano A, Suchindran S, Chisamore M, D'Souza JW, Faitg T, Rapoport AP. Safety and efficacy of letetresgene autoleucel alone or with pembrolizumab for relapsed/refractory multiple myeloma. Blood Adv. 2023 Apr 11;7(7):1168-1177. doi: 10.1182/bloodadvances.2022008460. PMID 36534160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a pilot study to assess safety and tolerability of genetically engineered New York esophageal squamous cell carcinoma 1 (NY-ESO-1) (c259) T Cells Alone or in combination with pembrolizumab in participants with relapsed/refractory multiple myeloma. The study was conducted in the United States.
Pre-assignment Details: A total of 127 participants were screened of which 6 participants were enrolled in the study. The study was terminated due to challenging screening and enrollment combined with a rapidly changing treatment landscape.
Groups:
- GSK3377794: Eligible participants underwent leukapheresis to manufacture engineered T-cells. Participants then underwent lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by a single intravenous (IV) infusion of GSK3377794.
- GSK3377794+Pembrolizumab: Eligible participants underwent leukapheresis to manufacture engineered T-cells. Participants then underwent lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by a single IV infusion of GSK3377794 in combination with pembrolizumab 200 milligrams (mg) administered as an IV infusion every 3 weeks up to Week 108.
Period: Overall Study
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
Started | 3 | 3
Completed | 3 | 2
Not Completed | 0 | 1
Not completed — Long term follow-up declined, study terminated by sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (11.27) | 64.3 (2.52) | 65.2 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant who received a study treatment and the event need not necessarily have a causal relationship with study treatment. An SAE is any AE that results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in a persistent or significant disability; is a congenital anomaly/birth defect; is clinically significant or requires intervention to prevent one of the outcomes listed before.
Time Frame: Up to 108 weeks
Population: Intent-To-Treat (ITT) Population comprised of all participants who underwent leukapheresis
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
Number analyzed (Participants) | 3 | 3
Participants
  Any AE | 3 | 3
  Any SAE | 2 | 2

2. Primary Outcome: Number of Participants With Treatment Limiting Toxicities-GSK3377794+Pembrolizumab Arm Only
Description: The following toxicities were considered to be treatment limiting toxicities: any >=Grade 4 AE; Grade 3 non-infectious pneumonitis and any other Grade 3 AE (excluding pneumonitis), that did not improve to Grade 2 within 7 days after onset despite medical management and supportive care. Exceptions included the following: Grade 3 or 4 leukopenia, lymphopenia, neutropenia, or febrile neutropenia; Grade 3 or 4 thrombocytopenia not associated with significant bleeding; Grade 3 anemia; Grade 4 cytokine release syndrome (CRS) or toxicities related to CRS that resolved to Grade <=2 within 7 days; other Grade 3 laboratory abnormality determined to be not clinically significant by the Investigator; Grade 3 or 4 fever and chills; Grade 3 or 4 hypoalbuminemia or abnormal electrolytes that responded to supplementation/correction; AE related to the cancer or its progression.
Time Frame: Up to 3 weeks
Population: ITT Population. Treatment limiting toxicities were assessed in GSK3377794+pembrolizumab arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3377794+Pembrolizumab
Number analyzed (Participants) | 3
Participants | 0

3. Primary Outcome: Number of Participants With Worst-case Chemistry Results by Any Grade Increase Post-Baseline Relative to Baseline
Description: Blood samples were collected for the assessment of following clinical chemistry parameters: glucose, albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, creatinine, potassium, magnesium, phosphate, sodium and calcium. Laboratory parameters were graded according to National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 4.03 where, Grade1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. An increase in grade is defined as an increase in CTCAE grade relative to Baseline grade. Data for any grade increase at worst case post Baseline is presented.
Time Frame: Up to 108 weeks
Population: Modified ITT Population comprised of all participants in the ITT Population who received the NY-ESO-1c259T infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
Number analyzed (Participants) | 3 | 3
Participants
  Glucose (Hyperglycemia) | 2 | 2
  Glucose (Hypoglycemia) | 0 | 0
  Albumin (Hypoalbuminemia) | 3 | 2
  ALP increased | 1 | 1
  ALT increased | 0 | 1
  AST increased | 0 | 1
  Bilirubin increased | 0 | 1
  Creatinine increased | 1 | 3
  Potassium (Hyperkalemia) | 0 | 0
  Potassium (Hypokalemia) | 1 | 2
  Magnesium (Hypermagnesemia) | 0 | 0
  Magnesium (Hypomagnesemia) | 2 | 1
  Phosphate (Hypophosphatemia) | 2 | 2
  Sodium (Hypernatremia) | 0 | 0
  Sodium (Hyponatremia) | 2 | 1
  Calcium (Hypercalcemia) | 1 | 0
  Calcium (Hypocalcemia) | 2 | 3

4. Primary Outcome: Number of Participants With Worst-case Hematology Results by Any Grade Increase Post-Baseline Relative to Baseline
Description: Blood samples were collected for the assessment of following hematology parameters: hemoglobin, lymphocytes, neutrophils, platelets and leukocytes. Laboratory parameters were graded according to NCI-CTCAE version 4.03 where, Grade1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. An increase in grade is defined as an increase in CTCAE grade relative to Baseline grade. Data for any grade increase at worst case post Baseline is presented.
Time Frame: Up to 108 weeks
Population: Modified ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
Number analyzed (Participants) | 3 | 3
Participants
  Hemoglobin (Anemia) | 2 | 3
  Hemoglobin increased | 0 | 0
  Lymphocyte count decreased | 3 | 3
  Lymphocyte count increased | 0 | 0
  Neutrophil count decreased | 3 | 3
  Platelet count decreased | 3 | 3
  Leukocyte count decreased | 3 | 3

5. Primary Outcome: Number of Participants With Worst-case Results for Coagulation Parameters Relative to Normal Range Post-Baseline Relative to Baseline
Description: Blood samples were collected for the assessment of following coagulation parameters: prothrombin time and partial thromboplastin time (PTT). A laboratory value that is outside the normal range is considered either high abnormal (value above the upper limit of the normal range) or low abnormal (value below the lower limit of the normal range). Participants were counted twice if the participant had values in 'Decreased to low' and 'Increased to high' during the post-Baseline period. Data for worst case post Baseline is presented.
Time Frame: Up to 108 weeks
Population: Modified ITT Population. Only those participants with data available at the specified time point is reported
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
Number analyzed (Participants) | 1 | 0
Participants
  Prothrombin Time; decrease to low | 0 |
  Prothrombin Time; To normal or no change | 0 |
  Prothrombin Time; increase to high | 1 |
  PTT; decrease to low | 0 |
  PTT; To normal or no change | 1 |
  PTT; increase to high | 0 |

6. Primary Outcome: Number of Participants With Worst-case Post Baseline Abnormal Electrocardiogram (ECG) Findings
Description: ECG was recorded using an ECG machine that automatically calculated the heart rate and measured PR, RR, QRS and QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals. Data for number of participants with abnormal clinically significant ECG findings for worst case post-Baseline has been presented. Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to 108 weeks
Population: Modified ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
Number analyzed (Participants) | 3 | 3
Participants | 0 | 1

7. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as the percentage of participants with a best overall response (BOR) of confirmed stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) per International Myeloma Working Group (IMWG) Response Criteria (2016); where, PR: >=50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by >=90% or to <200 milligrams (mg) per 24 hours; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours; CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <= 5% plasma cells in bone marrow; or sCR: CR as defined by normal free light chain (FLC) ratio and absence of clonal cells by immunohistochemistry. Confidence intervals were calculated using the exact (Clopper-Pearson) method.
Time Frame: Up to 108 weeks
Population: Modified ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
Number analyzed (Participants) | 3 | 3
Percentage of participants | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2]

8. Secondary Outcome: Time to Response
Description: Time to response is defined as the time interval (in months) from T-cell infusion to initial date of documented confirmed response (PR or better) in the subset of participants who showed a confirmed BOR of PR or better by Investigator assessment per IMWG (2016).
Time Frame: Up to 108 weeks
Population: Modified ITT Population. Only those participants with a confirmed response per IMWG 2016 were analyzed.
Measure: Median (Full Range); unit: Months
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
Number analyzed (Participants) | 1 | 2
Months | 0.7 [NA to NA] — Full range is not applicable as only a single participant was analyzed. Median value presented here is the actual time to response for this single participant. | 0.7 [0.7 to 0.7]

9. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the interval between the initial date of the confirmed response (sCR, CR, VGPR, or PR) and the initial assesment date of confirmed progressive disease or death among participants with a confirmed response per IMWG (2016).
Time Frame: Up to 108 weeks
Population: Modified ITT Population. Only those participants with a confirmed response per IMWG 2016 were analyzed.
Measure: Median (Full Range); unit: Months
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
Number analyzed (Participants) | 1 | 2
Months | 2.1 [NA to NA] — Full range is not applicable as only a single participant was analyzed. Median value presented here is the actual duration of response for this single participant. | 2.1 [2.1 to 2.1]

10. Secondary Outcome: Progression-free Survival
Description: Progression Free Survival is defined as the interval between the date of T-cell infusion and the initial assessment date of confirmed progressive disease as assessed by the investigator per IMWG (2016) or date of death. Progressive disease is defined as an increase of 25% from lowest confirmed response value in 1 or more of the following criteria: Serum M-protein with absolute increase of >=0.5 grams per deciliter (g/dL); Serum M-protein increase >=1 g/dL if the lowest M-component was >=5 g/dL; Urinary M-protein (absolute increase must be >=200 mg per 24 hours).
Time Frame: Up to 108 weeks
Population: Modified ITT Population
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
Number analyzed (Participants) | 3 | 3
Months | 2.79 [1.31 to 5.16] | 2.78 [2.76 to 2.79]

11. Secondary Outcome: Maximum Persistence (Cmax) of GSK3377794
Description: Blood samples were collected to measure persistence of infused GSK3377794 using polymerase chain reaction of a vector specific sequence in deoxyribonucleic acid (DNA) extracted from peripheral blood mononuclear cell (PBMC).
Time Frame: Up to 108 weeks
Population: Modified ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies per microgram genomic DNA
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
Number analyzed (Participants) | 3 | 3
Copies per microgram genomic DNA | 38509.67 (160.5) | 89640.56 (84.8)

12. Secondary Outcome: Time to Maximum Persistence
Description: Blood samples were collected to measure persistence of infused GSK3377794 using polymerase chain reaction of a vector specific sequence in DNA extracted from PBMC.
Time Frame: Up to 108 weeks
Population: Modified ITT Population
Measure: Median (Full Range); unit: Days
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
Number analyzed (Participants) | 3 | 3
Days | 8.0 [5 to 15] | 8.0 [7 to 15]

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Day 28 (AUC[0-28])
Description: as for outcome 12
Time Frame: Up to Day 28
Population: Modified ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days*Copies per microgram genomic DNA
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
Number analyzed (Participants) | 3 | 3
Days*Copies per microgram genomic DNA | 463989.35 (237.0) | 1498869.21 (90.4)

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected up to 108 weeks.
Description: Non-serious AEs and SAEs were collected in the ITT Population. All-cause mortality was collected in the modified ITT Population.
Arm/Group | GSK3377794 | GSK3377794+Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 2/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3377794 (N=3) | GSK3377794+Pembrolizumab (N=3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3377794 (N=3) | GSK3377794+Pembrolizumab (N=3)
Anaemia (Blood and lymphatic system disorders) | 3 (6) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (4) | 2 (2)
Fatigue (General disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 2 (3)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 2 (10) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (8) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood calcium increased (Investigations) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 2 (2)
Graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (7) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT03168438/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT03168438/SAP_001.pdf